CLINICAL TRIAL: NCT06188364
Title: Improving Traumatic Brain Injury Rehabilitation Care Transitions With Community Health Services: A Randomized Clinical Trial (CHW Intervention for TBI Care Transitions [CHWI for TBI]), a Research Project Within the TBI Model System
Brief Title: Improving Traumatic Brain Injury Rehab Care With Comm Health Services: a Research Project Within the TBI Model System
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20027800
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury
Keywords: Community Health Services; Rehabilitation Care Transitions; Caregiver Supports
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study is a single center, randomized clinical trial (RCT). We will use a block-randomization design with two arms:
  1. Usual Care Transition Supports and Services (USS) that prepare care partners of persons with TBI for post-rehabilitation discharge and
  2. Experimental USS supplemented with community health services delivered by a certified CHW (CHW+USS) for care partners:
     1. beginning within one week of inpatient rehabilitation discharge,
     2. active services (initiated by CHW or Care Partner) extending over 1- 12 weeks post-discharge, and
     3. passive services (initiated by care partner request only) 13-24 weeks post-discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): Transition Supports and Services (USS) that prepare care partners of persons with TBI for post-rehabilitation discharge
  Interventions: Other: Standard of Care
- Experimental (Experimental): USS supplemented with community health services delivered by a certified CHW (CHW+USS) for care partners
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Standard of Care — The usual Transition Supports and Services (USS) that prepare care partners of persons with TBI for post-rehabilitation discharge, so the the delivery of traditional CHW outreach services such as finding health, community and social determinants referrals, problem-solving, and connecting care partners to long-term supports/services
  Arms: Standard of Care
Other: Experimental — Novel aspects of the CHW experimental intervention for TBI care partners include:
  1. CHW services begin prior to inpatient rehabilitation discharge;
  2. care partners get timely, useful health management materials;
  3. encounters focus on unlimited, brief, situation-focused calls to help care partners assess and resolve pressing concerns; and
  4. long-term support capacity for care partners is built by establishing a reliable referral network of medical, community, and social services that become foundational resources beyond study completion.
  Arms: Experimental

SUMMARY:
TBI rehabilitation care transitions refer to the processes of preparing patients, families, and community-based healthcare providers for the patient's passage from inpatient rehabilitation to the home and community or to another level of care. Persons with TBI have heterogenous neurological impairment (cognitive and behavioral foremost, along with motor, sensory, and balance), that limits their functional independence and participation, and increases their risk for secondary medical conditions, injuries, rehospitalizations and early mortality

DETAILED DESCRIPTION:
Once people with TBI and their care partners enter the post-acute care landscape, they must navigate fragmented health care systems, interact with providers who may be unfamiliar with TBI, and discover their own services and supports. Inpatient rehabilitation provides high levels of structure and professional support that are impossible to replicate when constructing a home environment to independently manage day-to-day care. Once home, the person with TBI's physical, cognitive, behavioral, and medical needs can easily overwhelm even the most committed care partners. Community health workers (CHWs) through a combination of care coordination, advocacy, and direct service delivery, have the potential to address TBI care partners' needs, particularly those from low income and/or traditionally underserved minority groups. CHWs are well-suited to fill resource gaps that TBI care partners have difficulty finding, including: (1) finding diagnostic, treatment, and social services; (2) assisting with referrals; (3) providing health education and motivational interviewing to support behavioral health change; (4) collecting and managing clinical data; (5) facilitating productive relationships between health services and communities, and (6) offering psychosocial support.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults (age 18 or older).
* Must be primary person responsible for supervision/care needs of person with TBI post-IRF discharge.
* The person with TBI must have been admitted to the Brain Injury Service Unit at SAI.
* If the care partner does not live in the same residence as the person with TBI, they must provide multiple daily check-ins on day-to-day care.
* Must agree to use mHealth (texts, calls) and possess or be eligible to acquire a smart phone.

Exclusion Criteria:

* Any severe cognitive impairment that precludes the ability to provide informed consent or safely function as the care partner for a vulnerable adult with TBI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Managing Your loved Ones Health - Care Partner Activation | Measured at 12-weeks post-discharge
  Based on 32 self-report items prompt care partners to rate agreement with caregiving activity and engagement statements. Rated "1-Completely Agree" to "4-Completely Disagree" or "0 - Not My Responsibility."
  Used because:
  Good full-scale reliability (α=0.95). Sufficiently unidimensional for Rasch modeling with acceptable fit statistics, low standard error of measurement, and good range of item difficulty (23.8 - 71.8).
  Good concurrent validity: (a) positive correlations w/ care partner preparedness, self-competence, and self-confidence, and (b) negative correlations with stress, anxiety, and poor mental health

SECONDARY OUTCOMES:
Caregiver Well-Being Scale - Short Form (CWBS-SF) - Care Partner Well-Bing | Measured at 24-weeks post-discharge
  Based on 16 self-report items prompt care partners to rate representativeness of basic needs met and keeping up with day-to-day activities Rated from "1 - Rarely" to "5 - Usually."
  Used Because:
  Good full-scale reliability (α=0.83). Items have low redundancy; average inter-item r=.25 (range: .01 - .49). Good fit with two-factor model: (1) Basic Needs and (2) Implementation of Met Needs.
Patient Health Questionnaire - 4 (PHQ-4) - Care Partner Emotional Distress | Measured at 12- and 24-weeks post-discharge.
  Based on 4 self-report items prompt respondents to rate their depression and anxiety over last two weeks. Rated from "0 - Not at All" to "3 - Nearly Every Day."
  Used because:
  Good full-scale reliability (α=0.85). Clear 2-factor structure (anxiety and depression) explaining 84% of variance. High sensitivity as a screening scale.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Klyce, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States